CLINICAL TRIAL: NCT02830347
Title: Evaluation of the Changes in Oral and Gut Bacterial Resistance Caused by Short Term Antibiotic Treatment Following a Surgical Dental Procedure - A Prospective Clinical Study.
Brief Title: Changes in Resistome After Dental Extraction and Amoxicillin.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Michael G. Botelho, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: Version 1.1 (22.4.15)
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2016-07

CONDITIONS: Impacted Third Molar Tooth
Keywords: antibiotic resistance; oral microbiome
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
  Toungue coatings
  Stool samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Amoxicillin: No randomization is performed. Patients who are prescribed antibiotics by the clinician performing the tooth extraction ( based on case complexity and intra operative judgement) are recruited into this group.The principal investigator is not involved in the decision to prescribe antibiotics or not.
  Interventions: Drug: Amoxicillin; Procedure: Extraction
- No Amoxicillin: Patients who do not receive antibiotics after extractions are recruited into this group.
  Interventions: Procedure: Extraction

INTERVENTIONS:
Drug: Amoxicillin — Extraction
  Other Names: Aroxin
  Groups: Amoxicillin
Procedure: Extraction — Extraction of third molars

SUMMARY:
The aim of this study is to evaluate the nature of the change in oral and gut bacterial resistance profiles after antibiotic therapy for a surgical procedure in two groups. The intervention group will receive a course of amoxicillin and analgesics after surgical extraction and have bacterial samples taken from saliva, tongue coatings and stool samples at four appointments over a period of six months. This will be compared to the control group which receive only analgesics after the surgical extraction.

An examination of the development and sustainability of antibiotic resistance in the oral and gut microbiome of healthy cohorts will be followed up for 6 months, after surgical extraction of impacted teeth.

Change in proportion of antibiotic resistant bacterial components will be studied using Metagenomic DNA sequencing and quantification of resistant genes .

DETAILED DESCRIPTION:
Trial Design This is a prospective, longitudinal, observational, cohort study investigating young adults undergoing surgical extraction of a wisdom tooth with and without antibiotics post-operatively. The prescription of antibiotics will be based on clinical judgment based on case complexity, trauma and length of procedure. No randomization will be performed. Four observational time points will be undertaken for collecting 3 bacterial samples (tongue coating, saliva and stool sample at: baseline, 1 week, 1 month and 6 months.

To survey the extent and persistence of a range of bacterial resistance genes within the oral and gut microbiota of a cohort of systemically healthy young adults before and after the surgical extraction of third molars who receive and do not receive amoxicillin.

Hypothesis It is anticipated that a single course of amoxicillin (250 mg three times daily for five days) prescribed after a surgical tooth extraction, such as an impacted third molar, alters the short-term and long-term antibiotic resistance profile and causes a significant shift in the composition of the oral and gut resistome in a healthy cohort.

From analysis of the bacterial resistance, comparison from the baseline data over time will give insight on the impact of increased antibacterial resistance. Understanding of this should help pave the way for determining guidelines for the rational prescription of antibiotics for dental surgical clinical procedures and so form a basis for antibiotic stewardship as well as determine a potential risk to benefit awareness when prescribing antibiotics.

This baseline data can be followed-up in a longer timeframe to examine the persistence of resistance genes over time in a later study. It is expected a significant number of patients will be from student cohorts at HKU which will make later recall straightforward. Patients will be asked to keep a record log of antibiotic consumption after the initial study that may inform later research.

Subjects scheduled for surgical extractions who give a written consent to be a part of the study will be recruited. An experienced clinical operator with specialist maxillofacial surgery training (ML Co-A) will be responsible for performing clinical treatment. Prescription of antibiotics will be based on case complexity, difficulty of the operative surgical procedure and time taken. Therefore patients will not be randomized but based on obtaining 10 patients in each group. Three sets of samples (Saliva, tongue dorsum scrapings and stool samples) will be collected at the following four time points.

The subjects will be asked to refrain from brushing their teeth the night before sample collection is to be performed and similarly asked not to use dental mouthwashes. Apart from collection time points, subjects will be asked to maintain their 'normal', routine oral hygiene procedures for the duration of the study.

After collection of the baseline samples the surgical extraction of the third molar tooth will be performed. The subject will be given post extraction instructions and analgesics for pain relief for all the subjects and Amoxicillin for those requiring antibiotics. Compliance will be checked for by asking the patient and checking the tablet wrapper strips of amoxicillin at the recall appointments. The subject will be asked to refrain from using any mouth rinse during the six month study period (if they did not already do so) and a toothpaste without antibacterial content will be provided for use.

Tongue coating, saliva and stool samples for DNA extraction will be collected at all the specified time points as described below.

Baseline- antibiotic group On the day of surgery Baseline- no antibiotic On the day of surgery

1 week

1 week

1 month 6 months

Samples from the oral cavity will be taken in the morning at least two hours after meals. Subjects will be advised to collect the stool samples within 24 hours of the scheduled appointment.

A sterile micro brush will be used to collect the tongue coatings The tongue coating sample will be taken after stroking the surface of the tongue for three times from the back to the front side on one half of the anterior two-thirds of the tongue for each time point of sampling. After the sample collection, the tip of the micro brush will be cut and placed inside an Eppendorf vial. The samples will be stored at -800C until DNA extraction is performed.

For the saliva samples, the subject will be asked to spit out into a sterile container which will be immediately transferred into ice and then stored at - 800C. Collection of the stool samples will be performed based on the guidelines for stool sample collection given for the human microbiome project (16). DNA extraction will be performed from the samples using the DNA extraction kit provided by (Qiagen, USA).

Metagenomic shotgun sequencing For metagenomic sequencing extracted genomic DNA will be physically sheared to an average fragment size of 250 bp. The fragmented gDNA will be sequenced bi-directionally (100 bp each direction) on a lane of an Illumina HighSeq. Quality filtering will be performed with Trimmomatic (17), after which the paired and unpaired forward reads will be combined and reads with more than 10% ambiguous bases will be removed. Next, the reads will be screened for human sequences with Best Match Tagger v3.101 (18), after which human reads and duplicate reads will be removed.

Relative abundance of resistant genes The blaTEM primer used will be as described by Kim et al (22). Primers to analyze the presence of erm (G), erm (B) and erm (F) resistance genes will be as described by Jansonn et al (23). Primers for Tet (M) and Tet (W) genes will as described by Diaz-Torez et al (24). 16S universal primers will be used for the relative quantification as a standard.

12 The relative gene abundance will be assessed using real time PCR. Conventional PCR reactions will be used to generate gene-specific amplicons used as template DNA standards for qPCR. Amplicons will be purified using a gel/PCR extraction kit QIAquick PCR Purification Kit (Qiagen, USA) and quantified fluorometrically using a Quant-iTTM PicoGreen® dsDNA Assay Kit (Invitrogen). The number of DNA molecules will be calculated based on the size and mass of the amplicons. Tenfold serial dilutions of the amplicons will be prepared and used following the procedure by Yu et al. (25).

Selection and Withdrawal of Subjects Patients will be recruited from the waiting list from the Prince Philip Dental Hospital, The University of Hong Kong who have been clinically screened and wish to have their impacted wisdom teeth removed.

Sample size We would present the outcome in log 10 scale compared to day 0 in community DNA extracted from fecal samples. From the previous study (15), we anticipate the standard deviation as 1.25 units. By the sample size determination with the use of software G*Power version 3.1.9.2 (Franz Faul, Universitat Kiel, Germany), we would need at least 8 per group to have a power of 0.8 to detect the 1.25 unit difference at the 0.05 significance level. Therefore, in this research, we collect total sample size as 16 (8 per group) in the initial stage.

Treatment of Subjects This is a prospective, longitudinal, observational, cohort study investigating young adults undergoing surgical extraction of a wisdom tooth with and without antibiotics post-operatively. Antibiotics and analgesics will be given post- operatively.

Amoxicillin Intra orally, three times daily 250 mg for 5 days Analgesics - Arcoxia 120mg for three days and Paracetamol 500 mg QID PRN for 3 days or Paracetamol 1 g Plus 16 mg Codeine Phosphate. The prescription of antibiotics will be based on clinical judgment based on case complexity, trauma and length of procedure. No 14 randomization will be performed. Four observational time points will be undertaken for collecting 3 bacterial samples (tongue coating, mouth rinse and stool sample at: baseline, 1 week, 1 month and 6 months.

If the patients have to take additional antibiotics in the review period of six months, they will be asked to inform the investigator.

Compliance will be checked for by asking the patient and checking the tablet wrapper strips of amoxicillin at the recall appointments.

Assessment of Efficacy The study is not looking into the efficacy of a new drug. The treatment procedures being carried out are according to the conventional treatment protocol.

Assessment of Safety The study is not looking to the safety of a new drug. The treatment procedures being carried out are according to the conventional treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 45 years
2. Subjects who are scheduled to have a surgical tooth extraction.
3. Subjects who have signed an informed consent after being informed of the study design, objectives and, risks/benefits
4. No history of use of antibiotics up to three months prior to participation in the study.
5. No medical condition that prevents the surgical procedure or antibiotic therapy.
6. No history of hypersensitivity to beta lactams.
7. No contraindication to amoxicillin therapy.
8. Subjects are not pregnant or currently breast feeding.
9. No known or suspected immunodeficiency.

Exclusion Criteria:

1. History of antibiotic use within 3 months from baseline evaluation.
2. Any medical condition that prevents the surgical procedure or antibiotic therapy.
3. History of hypersensitivity to beta lactams
4. Contraindication for amoxicillin therapy
5. Pregnant or breast feeding women.
6. Subjects with known or suspected immunodeficiency.
7. Caries active subjects defined as subjects with active caries involving more than 3 teeth.
8. Subjects diagnosed with chronic periodontitis.
9. Subjects regularly using an antibacterial mouth rinse or planning to use one after the extraction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the waiting list from the Prince Philip Dental Hospital, Subjects scheduled for third molar extraction will be recruited based on the inclusion and exclusion criteria, provided they give a written informed consent for the acquisition of Saliva, tongue coatings and stool samples at the specified time points, after the study design and objectives have been explained in detail by the investigator.
  The prescription of antibiotics will be based on clinical judgment based on case complexity and the extent of the surgical trauma intra-operative Group 1- Surgical extraction with antibiotics-Amoxicillin 250 mg three times daily for 5 days and analgesics for pain relief.
  Group 2- Surgical extraction without antibiotics- Only analgesics for pain relief
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Quantification of antibiotic resistance genes by Resistance genes output at each timepoint from HUmanN 1.0 .Validation by QPCR values for Blatem and erm genes at each timepoint. | Baseline,One week,One month,Six months
  Resistome analysis Changes in the (relative) concentration of total resistance genes (the resistome) in the metagenomic DNA sequences will be analyzed as follows: Antibiotic resistance genes will be downloaded from the Antibiotic Resistance Genes Database (20). The downloaded dataset (ardbAnno1.0), containing 7828 entries, will be made non-redundant first and UBLAST from USEARCH v7.0.1090 (20) will be used to map the reads to the (ARDB) proteins (E-value threshold 10, post-filtered to include hits with a maximum E-value of 1E-10 inclusive).
  The results will be processed with HUMAN (21) to assign weights to the proteins. These weights were then normalized by dividing by the total number of filtered (non-human) reads, and summarized per antibiotic resistance type in the resistome. Next, fold changes will calculated for all resistance types with a baseline weight larger than 1E-8.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Botelho, BDS MSc PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Oral Rehabilitation, Faculty of Dentistry, The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data will be published within 6 months of the study completion.